CLINICAL TRIAL: NCT02046486
Title: OraL Crushed and dIspersed Ticagrelor 180mg Compared to Whole Tablets of eQUal Dose in STEMI Patients unDergoing Primary PCI: a Pharmacokinetic/Pharmacodynamic Study
Brief Title: OraL Crushed and dIspersed Ticagrelor 180mg Compared to Whole Tablets of eQUal Dose in STEMI Patients unDergoing Primary PCI: a Pharmacokinetic/Pharmacodynamic Study (the LIQUID Study)
Acronym: LIQUID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIQUID study
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ticagrelor; ST elevation myocardial infarction; liquid formulation
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor 180mg whole tablets (Active Comparator): Ticagrelor 180mg loading dose, in the form of 2 whole tablets administered per os in the supine position (standard administration)
  Interventions: Drug: Ticagrelor 180mg whole tablets
- Ticagrelor 180mg crushed and dispersed (Experimental): Ticagrelor 180mg in the form of 2 tablets crushed and dispersed in purified water administered per os with 1-minute-stay in a 60-70 degrees semi-upright sitting position
  Interventions: Drug: Ticagrelor 180mg crushed and dispersed

INTERVENTIONS:
Drug: Ticagrelor 180mg whole tablets
  Arms: Ticagrelor 180mg whole tablets
Drug: Ticagrelor 180mg crushed and dispersed
  Arms: Ticagrelor 180mg crushed and dispersed

SUMMARY:
This is a single-center, prospective, randomized, single-blind, investigator initiated, pharmacokinetic/pharmacodynamic study of parallel design.Patients with ST elevation myocardial infarction (symptom onset<12 hours), undergoing primary percutaneous coronary intervention, who are P2Y12 inhibitor naïve, will be randomized after informed consent, immediately after diagnostic coronary angiography, in a 1:1 ratio to either:

* Ticagrelor 180mg loading dose, in the form of 2 whole tablets administered per os in the supine position (standard administration)
* Ticagrelor 180mg loading dose, in the form of 2 tablets crushed and dispersed in purified water and administered per os with 1-minute-stay in a 60-70 degrees semi-upright sitting position Platelet reactivity assessment will be performed at randomization (Hour 0) and at 0.5, 1, 2, 4 and 6 hours after randomization, using the VerifyNow assay, in platelet reactivity units (PRU). The cutoff >208 PRU will be used for definition of high platelet reactivity (HPR). All platelet reactivity assessments will be performed by a physician blind to the actual treatment given. Additional blood samples will be collected at the same time points for pharmacokinetic analysis. These samples will be collected in vacuum tubes with lithium heparin and will be kept in ice until centrifugation (3000 rpm at 4°C for 10 min, within 30 min of sampling). The resultant plasma will be transferred into a plain polypropylene tube (screw cap) and stored at or below -20°C until analysed.

DETAILED DESCRIPTION:
Preparation of Ticagrelor liquid formulation:

Crushed and dispersed Ticagrelor 180mg for oral administration will be prepared as follows: two ticagrelor 90mg tablets are placed in a mortar and crushed for 60 s using a pestle. 20 mL of purified water will be added in the mortar and stirred for 60s. The liquid is transferred to a dosing cup and another 15 mL of purified water is added to the mortar and stirred, ensuring that all powder has been dispersed and none remained on the mortar and pestle. Again the liquid is transferred to the dosing cup. The same procedure is repeated with 15 ml of purified water.The total contents are stirred for another 30 s to ensure that all remaining tablet particles are dispersed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients with STEMI (onset of pain<12 hours) with indication for primary PCI
3. Informed consent obtained in writing

Exclusion Criteria:

Pregnancy/Breastfeeding

* Severe nausea or vomiting
* Treatment with a P2Y12 inhibitor within the previous 1 month
* Inability to give informed consent
* Hemodynamic instability
* Arrhythmias requiring cardioversion, temporary pacemaker insertion or intravenous antiarrhythmic agents
* Killip class ≥3
* Known hypersensitivity to ticagrelor
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding
* Thombocytopenia (<100.000 / μL) at randomization
* Anaemia (Hct <30%) at randomization
* Polycytaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitor administration
* Thrombolysis administration
* Recent (< 6 weeks) major surgery or trauma, including GABG.
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine).
* Patients considered by the investigator to be at increased risk of bradycardiac events.
* Dialysis required.
* Severe uncontrolled chronic obstructive pulmonary disease
* Known severe hepatic impairement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Ticagrelor's Cmax over 1 hour post ticagrelor administration | 1 hour
Area under the ticagrelor plasma concentration versus time curve (AUC0-1) over 1 hour post ticagrelor administration | 1 hour

SECONDARY OUTCOMES:
Platelet reactivity at 1 hour post randomization | 1 hour
  Platelet reactivity assessment with the VerifyNow assay
HPR rate at 1 hour post randomization | 1 hour
  HPR rate at 1 hour post randomization between the two treatment arms
Platelet reactivity at 2 hours post randomization | 2 hours
  Platelet reactivity assessment with the VerifyNow assay
HPR rate at 2 hours post randomization | 2 hours
  HPR rate at 2 hours post randomization between the 2 treatment arms.
AR-C124910XX Cmax over 1 hour post ticagrelor administration | 1 hour
AR-C124910XX Cmax over 6 hours post ticagrelor administration | 6 hours
Ticagrelor Cmax over 6 hours post ticagrelor administration | 6 hours
Area under the AR-C124910XX plasma concentration versus time curve (AUC0-1) over 1 hour post ticagrelor administration | 1 hour
Area under the AR-C124910XX plasma concentration versus time curve (AUC0-6) over 6 hours post ticagrelor administration | 6 hours
Area under the Ticagrelor plasma concentration versus time curve (AUC0-6) over 6 hours post ticagrelor administration | 6 hours
Time for the maximum plasma concentration (Tmax) of Ticagrelor over 6 hours post Ticagrelor administration | 6 hours
Time for the maximum plasma concentration (Tmax) of AR-C124910XX over 6 hours post Ticagrelor administration | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital Department of Cardiology, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Alexopoulos D, Barampoutis N, Gkizas V, Vogiatzi C, Tsigkas G, Koutsogiannis N, Davlouros P, Hahalis G, Nylander S, Parodi G, Xanthopoulou I. Crushed Versus Integral Tablets of Ticagrelor in ST-Segment Elevation Myocardial Infarction Patients: A Randomized Pharmacokinetic/Pharmacodynamic Study. Clin Pharmacokinet. 2016 Mar;55(3):359-67. doi: 10.1007/s40262-015-0320-0. PMID 26315810